CLINICAL TRIAL: NCT05876117
Title: Clonidine and Lorazepam Premedication for Claustrophobic Patients During MRI Scan
Brief Title: Premedication for Claustrophobic Patients for MRI Scan
Status: Recruiting | Type: Observational
Sponsor: Salem Anaesthesia Pain Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: SalemAnes2022 MRI Premedicate
Record Dates: First submitted 2023-05-05; First posted 2023-05-25 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Claustrophobia
Keywords: Claustrophobia MRI
MeSH Terms: conditions — Claustrophobia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Claustrophobic adult patients: Claustrophobic adult patients who are undergoing MRI scan as part of chronic pain management.

SUMMARY:
Claustrophobia is an irrational fear of restriction and suffocation. It is a specific phobia, according to DSM 5. Claustrophobic patients may fear that restriction of their limbs will hinder their ability to move quickly towards safety. MRI may trigger claustrophobia, because this diagnostic procedure involves a patient laying in a narrow tube. Premedication before MRI scan may occasionally reduce claustrophobia.

Prospective observational crossover study of claustrophobic patients who are undergoing MRI scan. At alternate MRI scan sessions, each patient receives rotational premedication using Lorazepam 1mg; or Clonidine tablet 0.2mg; or combined Clonidine 0.2mg + Lorazepam 1mg.

Patient will use Claustrophobia Questionnaire, a validated tool, to collect data on the days before and after each MRI scan. CLQ is a patient-administered tool used to assess claustrophobia. In addition, patient will use General Anxiety Disorder Questionnaire, a validated tool, to collect data on the days before and after each MRI scan. GAD-7 is a patient-administered tool that is used to assess anxiety.

DETAILED DESCRIPTION:
Claustrophobia is an irrational fear of constraint, restriction, immobility, smothering and suffocation. Claustrophobia is a specific phobia, according to the Diagnostic and Statistical Manual 5 (DSM 5). The disorder affects 5% of the general population. Claustrophobic patients may fear that the restriction of their limbs will hinder their ability to move quickly towards perceived safety. Magnetic resonance imaging (MRI) may trigger claustrophobia, because this diagnostic procedure involves a patient staying immobile in a narrow and noisy tube. Anxiolytic premedication before MRI scan, using Lorazepam, may occasionally help to reduce claustrophobia.

This is a prospective observational crossover study of claustrophobic adult patients who are undergoing MRI scan as part of chronic pain management. At alternate MRI scan sessions, each patient receives rotational premedication using Lorazepam 1mg; or Clonidine tablet 0.2mg; or combined Clonidine 0.2mg + Lorazepam 1mg.

The patient will use the Claustrophobia Questionnaire (CLQ), a special validated tool, to collect data on the days before and after each MRI scan. The CLQ is a patient-administered tool that is used to record the severity and presence of claustrophobia symptoms, on a measurement range of 0 to 104. A change in the CLQ scores by 12-points is considered significant. In addition, the patient will use the General Anxiety Disorder Questionnaire (GAD-7), a special validated tool, to collect data on the days before and after each MRI scan. The GAD-7 is a patient-administered tool that is used to record the severity and presence of anxiety symptoms, on a measurement range of 0 to 21. A change in the GAD-7 scores by 3-points is considered significant.

Data analyzed with IBM® SPSS® Statistics 25 (IBM Corp, Armonk, NY); using Student's t-test, ANOVA, Pearson Chi-square test, and regression analysis. P-value <0.05 is considered significant.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with claustrophobia
* previous incomplete MRI because of claustrophobia
* adult patients
* good treatment compliance
* reliable Claustrophobia Questionnaire (CLQ) diary
* reliable General Anxiety Disorder Questionnaire (GAD) diary
* informed consent for diary review
* consent for clinical record quality assurance review

Exclusion Criteria:

* poor treatment compliance
* cognitive disorder
* inability to provide consent
* major neuropsychiatric disorder
* unreliable diary
* cannabis use
* excessive alcohol intake
* previous adverse/allergic reactions to clonidine
* previous adverse/allergic reactions to lorazepam

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult claustrophobic patients who are undergoing MRI scan as part of chronic pain management. Previous incomplete MRI because of claustrophobia.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-07-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of completion of MRI scan | 12 weeks
  Patient is calm and cooperative, completes MRI scan

CONTACTS AND LOCATIONS:
Overall Officials: Olu Bamgbade, MD,FRCPC, Principal Investigator — Salem Anaesthesia Pain Clinic
Locations (1):
- Salem Anaesthesia Pain Clinic, Surrey, British Columbia, Canada